CLINICAL TRIAL: NCT05866718
Title: Can Applying the Science of Habit Formation to Contemplative Practice Improve Outcomes? A Randomized Controlled Trial of a Single-Session Habit Formation Intervention for Self-Compassionate Touch
Brief Title: Can Applying the Science of Habit Formation to Contemplative Practice Improve Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other); The Greater Good Science Center at the University of California, Berkeley (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-12-14924-2
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Psychopathology
Keywords: Self-Compassion; Single-Session Intervention; Transdiagnostic; Intervention; Habits; Habit Formation; Micropractice; Contemplative Micropractice; Contemplative Practice; Self-Compassionate Touch; Compassion
MeSH Terms: conditions — Habits

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the SCT or SCT+HABITS using the randomizer elements in Qualtrics.
Who Masked: Participant
Masking Description: Study participants will not be made aware that there are two experimental conditions. All will be told that they are receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassionate Touch Intervention Alone (Active Comparator): All participants will receive the self-compassion intervention after completing their baseline assessment, which will contain the same instructions used in the initial study (see NCT05199779).
  Interventions: Behavioral: Self-Compassionate Touch Intervention
- Self-Compassionate Touch Intervention Plus Habit Formation Tools (Experimental): SCT+HABITS participants will receive the abovementioned procedures, and will also receive evidence-based tools for forming habits.
  Interventions: Behavioral: Self-Compassionate Touch Intervention; Behavioral: Habit Formation Tools

INTERVENTIONS:
Behavioral: Self-Compassionate Touch Intervention — Participants will be taught the micropractice (<20-second/day personal practice) via video recording.
Behavioral: Habit Formation Tools — Participants will receive evidence-based tools for promoting habit-formation.
  Arms: Self-Compassionate Touch Intervention Plus Habit Formation Tools

SUMMARY:
In the present study, the investigators will conduct a confirmatory efficacy trial to test whether improving practice automaticity (i.e., habit formation) of self-compassionate touch improves outcomes in the predicted direction. Adults (n=440, including 20% for attrition) will be randomly assigned to: (1) the self-compassionate touch intervention plus habit formation tools ("SCT+HABITS") versus (2) the self-compassionate touch intervention alone ("SCT"). The investigators will conduct assessments at baseline, 3-month follow-up, and 6-month follow-up. The SCT+HABITS condition will be used to evaluate whether providing habit formation tools results in superior effects to SCT. The intervention will be delivered entirely online.

DETAILED DESCRIPTION:
Specific Aim 1: Evaluate whether SCT+HABITS shows more practice frequency and practice automaticity from baseline to 3-month, and to 6-month follow-up compared to the SCT. Hypothesis 1. The SCT+HABITS group will show greater increases in practice frequency and practice automaticity than SCT from baseline to 3-month, and to 6-month follow-up.

Specific Aim 2: Determine whether SCT+HABITS, relative to SCT, will experience increased self-compassion and self-compassion automaticity, and reduced stress and psychopathology. Hypothesis 2. SCT+HABITS will promote greater increases in self-compassion and self-compassion automaticity, and greater reductions in stress and psychopathology from baseline to 3-month, to 6-month follow-up.

Specific Aim 3: Assess whether greater baseline to 3-month follow-up increases in practice automaticity mediate the association between SCT+HABITS and baseline to 6-month follow-up increases in (a) self-compassion and (b) self-compassion automaticity, as well as reductions in (c) stress and (d) psychopathology. Hypothesis 3. Greater baseline to 3-month follow-up increases in practice automaticity will mediate the association between the SCT+HABITS group and baseline to 6-month follow-up increases in (a) self-compassion and (b) self-compassion automaticity, as well as reductions in (c) stress and (d) psychopathology.

Exploratory Aim: Evaluate the barriers, facilitators, and acceptability of SCT+HABITS and SCT alone. This aim will be addressed via qualitative analyses to characterize barriers and facilitators to habit formation, and the proportion of participants in each condition (SCT+HABITS and SCT alone) who noted each type of barrier and facilitator. Participants will self-report on acceptability and feasibility via questionnaire. Then, the investigators will examine whether SCT+HABITS and SCT alone will meet or exceed the established criteria for acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* English language proficiency.
* Able and willing to give informed consent.
* Resides in the United States of America

Exclusion Criteria:

* Does not have email address or access to email.
* Does not personally own a smartphone device
* Not able/willing to participate in and/or complete the baseline assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-09-22 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
Practice Frequency | Change from baseline to 3-month follow-up, and to 6-month followup
  Number of times practiced self-compassion exercise per week since last assessment. 1 item. Higher frequency indicates a better outcome.
Practice Automaticity (Practice Self-Report Behavioral Automaticity Index [SRBAI]) | Change from baseline to 3-month follow-up, and to 6-month follow-up.
  4 items, 1-9 scale. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Self-Compassion (Sussex-Oxford Compassion for the Self Scale [SOCS-S]) | Change from baseline to 3-month follow-up, and to 6-month followup
  20-items, 5-point response scale. Scores can range from 20 to 100 (Higher score means higher compassion for self). Sub-scale items included.
Self-Compassion Automaticity (Self-Compassion Self-Report Behavioral Automaticity Index [SRBAI]) | Change from baseline to 3-month follow-up, and to 6-month followup.
  20 items. 1-9 scale. Higher scores indicate a better outcome.
Perceived Stress (Perceived-Stress Scale [PSS-10]) | Change from baseline to 3-month follow-up, and to 6-month followup
  10 items, 5 point response scale (from 0 = Never to 4 = Very Often). Lower scores indicate a better outcome.
  Scoring: Reverse score (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) items 4, 5, 7, & 8 and then summing across all scale items.
Psychopathology (DSM-5 Cross-Cutting Measure [DSM-XC]) | Change from baseline to 3-month follow-up, and to 6-month followup
  22 items (suicidality item Q11 removed). 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day).

OTHER OUTCOMES:
Barriers and Facilitators | Assessed at 6-month followup
  The investigators will explore first-person experience of using the practice by asking open-ended free-response questions. The investigators will develop a coding system of the barriers and facilitators to forming the habit of practicing SCT daily.
Acceptability and Feasibility (Program Feedback Scale [PFS]) | Assessed at 6-month followup
  7 Items. 5-point scale (1="really disagree"; 5="totally agree")

CONTACTS AND LOCATIONS:
Overall Officials: Eli S Susman, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California at Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the Open Science Framework by time of publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared via the Open Science Framework by time of publication.
Access Criteria: De-identified data, materials and analytic code will be made publicly available